CLINICAL TRIAL: NCT05383274
Title: Optilume PoST AppRoval Clinical Evaluation of Andrology ParaMeters
Acronym: STREAM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Urotronic Inc. (Industry)
Collaborators: Laborie Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR1275
Record Dates: First submitted 2022-05-16; First posted 2022-05-20 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Urethral Stricture
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Optilume Urethral DCB (Experimental): The Optilume Drug Coated Balloon (DCB) is a guidewire compatible catheter with a tapered atraumatic tip. The distal end of the catheter has an inflatable balloon coated with a proprietary coating containing the drug paclitaxel that facilitates the drug's transfer to the urethral wall upon inflation.
  Interventions: Combination Product: Optilume Urethral DCB

INTERVENTIONS:
Combination Product: Optilume Urethral DCB — The Optilume Drug Coated Balloon (DCB) is a guidewire compatible catheter with a tapered atraumatic tip. The distal end of the catheter has an inflatable balloon coated with a proprietary coating containing the drug paclitaxel that facilitates the drug's transfer to the urethral wall upon inflation.

SUMMARY:
Single-arm, prospective study assessing semen quality after treatment with the Optilume Urethral DCB in men between 22 and 65 years of age.

DETAILED DESCRIPTION:
Male subject diagnosed with a stricture in the anterior urethra that can be treated with the Optilume Urethral DCB. Thirty-Four (34) subjects will be enrolled at up to ten (10) sites in the United States. Clinical follow-up will be conducted at 30 days, 3 months, 6 months, and 12 months post-treatment evaluating Lower Urinary Tract Symptoms (LUTS), sexual function, and voiding function. Semen quality parameters will be assessed at Baseline, 3 months, and 6 months post-treatment. Subjects with an abnormal semen quality result at 6 months will have an additional assessment at 12 months post-treatment and periodically thereafter until results return to normal.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects between 22 and 65 years of age
2. Subject diagnosed with a stricture in the anterior urethra that is able to be treated with the Optilume Urethral DCB in accordance with the approved Instructions for Use
3. Subject is willing to provide written informed consent and comply with study required follow-up assessments
4. Subject able to provide viable semen samples and baseline semen quality characteristics are above reference values based on below criteria (average of 2 samples):

   1. total sperm ≥39 million
   2. sperm concentration ≥15 million/mL
   3. total motility ≥40%
   4. progressive motility ≥32%
   5. morphology ≥4%

Exclusion Criteria:

1. Subjects with a known hypersensitivity to paclitaxel or structurally related compounds
2. Subjects with a history of vasectomy or other condition that may inhibit semen/sperm production or ejaculatory function
3. Subjects currently taking 5-alpha reductase inhibitors, alpha-blockers, selective serotonin reuptake inhibitors, or hormone replacement therapy without appropriate washout
4. Subject is unwilling to abstain or utilize a condom for 30 days after the procedure
5. Subject is unwilling to utilize highly effective contraception for 6 months after the procedure if partner is of childbearing potential
6. History of cancer in any body system that is not considered in complete remission

Ages: 22 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men between 22 and 65 years of age.
Enrollment: 34 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 3-months
  Average Change in Sperm Concentration from baseline to 3-months

SECONDARY OUTCOMES:
Secondary Safety Endpoint | 6-months
  Proportion of Subjects Experiencing ≥50% Decrease in Sperm Concentration from Baseline at 3 and 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Karl Coutinho, MD, Principal Investigator — New Jersey Urology
Locations (9):
- United States (9):
  - Arkansas Urology, Little Rock, Arkansas
  - Orlando Health, Orlando, Florida
  - Florida Urology, Tampa, Florida
  - Regional Urology, Shreveport, Louisiana
  - Chesapeake, Hanover, Maryland
  - Freedman Urology, Las Vegas, Nevada
  - New Jersey Urolgy, Millburn, New Jersey
  - Western New York, Cheektowaga, New York
  - Urology Clinics of North Texas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No